CLINICAL TRIAL: NCT01974167
Title: Eldecalcitol for GLucocorticoid Induced OsteopoRosIs Versus Alfacalcidol
Acronym: e-GLORIA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: e-GLORIA trial Protocol Review Committee (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013/9/9 Ver1.0; UMIN000011700 (Registry Identifier: UMIN)
Record Dates: First submitted 2013-10-28; First posted 2013-11-01 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-05

CONDITIONS: Osteoporosis
Keywords: glucocorticoid-induced osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — eldecalcitol; alfacalcidol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eldecalcitol group (Experimental): Eldecalcitol 0.75 microgram once daily orally
  Interventions: Drug: Eldecalcitol
- Alfacalcidol group (Active Comparator): Alfacalcidol 1 microgram once daily orally
  Interventions: Drug: Alfacalcidol

INTERVENTIONS:
Drug: Eldecalcitol — Eldecalcitol 0.75 microgram once daily orally
  Arms: Eldecalcitol group
Drug: Alfacalcidol — Alfacalcidol 1 microgram once daily orally
  Arms: Alfacalcidol group

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of eldecalcitol monotherapy compared with alfacalcidol monotherapy in patients with glucocorticoid-induced osteoporosis, using a randomized, open-label, parallel-group, comparative design.

ELIGIBILITY:
Inclusion Criteria:

* (1) Patients who are currently taking or plan to take oral glucocorticoid medication for 3 months or longer and thus require treatment as per the 'Guidelines on the management and treatment of glucocorticoid-induced osteoporosis of the Japanese Society for Bone and mineral Research (2004),' and who meet at least one of the conditions below. No restriction is imposed on the underlying disease treated with the oral glucocorticoid medication.

  (i) Have any existing insufficiency fracture (ii) %YAM <80 (iii) Oral glucocorticoid daily dose >= 5 mg prednisolone equivalent
* (2) Aged between 20 and 85 years (both inclusive) at consent
* (3) Patients who are able to walk without assistance
* (4) Provided consent to participate in the study

Exclusion Criteria:

* (1) BMD (L1-4 or T-Hip) T score < -3.5
* (2) Have 3 or more vertebral fractures between L1 and L4.
* (3) Have 1 or more SQ grade 3 vertebral fractures, or 3 or more SQ grade 2 vertebral fractures.
* (4) Have received a bisphosphonate preparation for 2 weeks or longer within 6 months before the start of study treatment.
* (5) Have received a bisphosphonate preparation for 2 years or longer within 3 years before the start of study treatment.
* (6) Have received a parathyroid hormone preparation before the start of study treatment.
* (7) Have received one or more doses of an anti-RANKL (receptor activator of nuclear factor-kappa B ligand) antibody.
* (8) Have received one or more doses of an anti-sclerostin antibody or cathepsin K inhibitor.
* (9) Have received any other investigational product (including placebo) within 16 weeks before the start of study treatment in the present study.
* (10) Have received any of the following drugs that can affect bone metabolism within 8 weeks before the start of study treatment, with the exception of calcium preparations: (i) Bisphosphonates (ii) Active vitamin D preparations (including those for topical use) (iii) Selective estrogen receptor modulators (SERMs) (iv) Calcitonin preparations (v) Vitamin K2 preparations (vi) Ipriflavone preparations (vii) Reproductive hormone products (except those for vaginal use such as vaginal tablets and creams) (viii) Other drugs that can affect bone metabolism
* (11) Pregnant woman or woman who desires to become pregnant
* (12) Have corrected serum calcium >= 10.4 mg/dL or < 8.0 mg/dL at enrollment.
* (13) Have corrected urinary calcium > 0.4 mg/dL GF at enrollment.
* (14) Have a past or current history of urinary calculus.
* (15) Have eGFR < 30 mL/min/1.73 m2 at enrollment.
* (16) Have severe liver disease such as cirrhosis or severe heart disease such as severe cardiac failure.
* (17) Have active malignancy or received treatment for malignancy, including adjuvant therapy, within the past 3 years.
* (18) Have a history of hypersensitivity to eldecalcitol, alfacalcidol, or other vitamin D preparations.
* (19) Other persons judged by the investigator (or subinvestigator) to be inappropriate to participate in this study.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2013-12; Primary Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Percent change in lumbar spine (L1-4) bone mineral density | 12 months after the start of study drug administration
Incidence of vertebral fractures | 36 months
  A vertebral fracture will be classified as a new fracture (i.e., change from grade 0 to grade 1, 2, or 3) or worsening of a prevalent fracture (i.e., change from grade 1 to grade 2 or 3, or change from grade 2 to grade 3) using a semi-quantitative [SQ] method according to the "Vertebral Fracture Assessment Criteria, 2012 revised version."

SECONDARY OUTCOMES:
Incidence of non-vertebral fractures (both traumatic and non-traumatic; All sites) | 36 months
Incidence of non-vertebral fractures (both traumatic and non-traumatic; 3 Major sites) | 36 months
  The 3 Major sites are defined as the forearm, humerus, and femur.
Incidence of non-vertebral fractures (both traumatic and non-traumatic; 6 Major sites) | 36 months
  The 6 Major sites are defined as the femur, lower leg, humerus, forearm, clavicle, and pelvis.
Incidence of non-vertebral fractures (traumatic; All sites) | 36 months
Incidence of non-vertebral fractures (traumatic; 3 Major sites) | 36 months
Incidence of non-vertebral fractures (traumatic; 6 Major sites) | 36 months
Incidence of non-vertebral fractures (non-traumatic; All sites) | 36 months
Incidence of non-vertebral fractures (non-traumatic; 3 Major sites） | 36 months
Incidence of non-vertebral fractures (non-traumatic; 6 Major sites） | 36 months
Incidence of vertebral fractures (new vertebral fractures) | 36 months
Incidence of vertebral fractures (worsening of prevalent vertebral fractures) | 36 months
Incidence of vertebral fractures (clinical vertebral fractures) | 36 months
Incidence of vertebral fracture (new or worsening of prevalent fractures) by glucocorticoid dose | 36 months
Incidence of clinical vertebral fractures by glucocorticoid dose | 36 months
Incidence of non-vertebral fractures (all sites) by glucocorticoid dose | 36 months
Incidence of non-vertebral fractures (3 Major sites) by glucocorticoid dose | 36 months
Incidence of non-vertebral fractures (6 Major sites) by glucocorticoid dose | 36 months
Incidence of vertebral fractures (new or worsening) by bone mineral density | 36 months
Incidence of clinical vertebral fractures by bone mineral density | 36 months
Incidence of non-vertebral fractures (all sites) by bone mineral density | 36 months
Incidence of non-vertebral fractures (3 Major sites) by bone mineral density | 36 months
Incidence of non-vertebral fractures (6 Major sites) by bone mineral density | 36 months
Incidence of vertebral fractures (new or worsening) by number of prevalent fractures | 36 months
Incidence of clinical vertebral fractures by number of prevalent fractures | 36 months
Incidence of non-vertebral fractures (all sites) by number of prevalent fractures | 36 months
Incidence of non-vertebral fractures (3 Major sites) by number of prevalent fractures | 36 months
Incidence of non-vertebral fractures (6 Major sites) by number of prevalent fractures | 36 months
Incidence of new vertebral fractures by severity | 36 months
  Semiquantitative (SQ) method is used for grading of vertebral fractures.
Incidence of new clinical vertebral fractures by severity | 36 months
  SQ method is used for grading of vertebral fractures.
Incidence of new non-vertebral fractures (all sites) by severity | 36 months
  SQ method is used for grading of vertebral fractures.
Incidence of new non-vertebral fractures (3 Major sites) by severity | 36 months
  SQ method is used for grading of vertebral fractures.
Incidence of new non-vertebral fractures (6 Major sites) by severity | 36 months
Incidence of osteoporotic fractures | 36 months
  An osteoporotic fracture is defined as a fracture of the following sites: vertebral body, ribs, pelvis, humerus, clavicle, scapula, sternum, proximal femur, other portions of the femur, tibia, fibula, and forearm.
Incidence of FRAX-defined major osteoporotic fractures | 36 months
  The 4 Major sites are defined as clinical fractures of the spine, forearm, hip, and shoulder.
Percent change in lumbar spine bone mineral density | 6 months after the start of study drug administration
Percent change in lumbar spine bone mineral density | 24 months after the start of study drug administration
Percent change in lumbar spine bone mineral density | 36 months after the start of study drug administration (or at the time of withdrawal from the study)
Change in proximal femur (total-hip) bone mineral density | 6 months after the start of study drug administration
Change in proximal femur (total-hip) bone mineral density | 12 months after the start of study drug administration
Change in proximal femur (total-hip) bone mineral density | 24 months after the start of study drug administration
Change in proximal femur (total-hip) bone mineral density | 36 months after the start of study drug administration (or at the time of withdrawal from the study)
Percent change in TRACP-5b bone metabolism marker | 6 months after the start of study drug administration
Percent change in TRACP-5b bone metabolism marker | 12 months after the start of study drug administration
Percent change in PINP bone metabolism marker | 6 months after the start of study drug administration
Percent change in PINP bone metabolism marker | 12 months after the start of study drug administration
Frequency of falls | 36 months
Change in muscle strength (back muscle strength) | 12 months after the start of study drug administration
Change in muscle strength (back muscle strength) | 24 months after the start of study drug administration
Change in muscle strength (back muscle strength) | 36 months after the start of study drug administration (or at the time of withdrawal from the study)
Change in muscle strength (grip strength) | 12 months after the start of study drug administration
Change in muscle strength (grip strength) | 24 months after the start of study drug administration
Change in muscle strength (grip strength) | 36 months after the start of study drug administration (or at the time of withdrawal from the study)
Change in height | 12 months after the start of study drug administration
Change in height | 24 months after the start of study drug administration
Change in height | 36 months after the start of study drug administration (or at the time of withdrawal from the study)

CONTACTS AND LOCATIONS:
Overall Officials: Toshio Matsumoto, Study Chair — University of Tokushima
Locations (1):
- Nara Hospital Kinki University Faculty of Medicine, Ikoma, Nara, Japan